CLINICAL TRIAL: NCT06603168
Title: Autonomic Recalibration Approach to Myofascial Pain Elimination
Brief Title: Autonomic Recalibration
Acronym: ART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Edward Via Virginia College of Osteopathic Medicine (Other)
Responsible Party: Principal Investigator, William Pearson, Discipline Chair for Anatomy, Edward Via Virginia College of Osteopathic Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-058
Record Dates: First submitted 2024-09-17; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Chronic Pain (Back / Neck); Autonomic Dysregulation
Keywords: chronic pain; autonomic nervous system; sympathetic dominance; myofascial pain; Sympathetic tone; dysfunctional pain; Primal Reflex Release Technique; shear wave elastography; heart rate variability; galvanic skin response; Rokoko; motion capture; range of motion; posture
MeSH Terms: conditions — Chronic Pain; Primary Dysautonomias

STUDY DESIGN:
Intervention Model Description: This pilot study design is a pretest-posttest cohort study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Autonomic Recalibration Treatment (Experimental): Participant receives Autonomic Recalibration Treatment.
  Measurements:
  Pre/post shear wave elastography Pre/post myonometry Pre/post motion capture HRV/GSR during ART Pre/post pain ratings Pre/post trigger point log
  Interventions: Other: Autonomic Recalibration Treatment

INTERVENTIONS:
Other: Autonomic Recalibration Treatment — An initial history to r/o pathology and document a chief complaint relevant to pain is conducted. An initial head to toe assessment of withdrawal or startle reflex behavior in response to palpation is performed to identify trigger points and establish patterns of sympathetic dominance throughout the myofascial system. The pattern of sympathetic dominance (pattern of trigger point) is addressed during treatment by Primal Reflex Release Technique Protocol to inhibit somatic afferent feedback loops and rebalance the autonomic nervous system towards a state of parasympathetic dominance. The absence of a trigger point indicates that the treatment is complete.

SUMMARY:
The goal of this clinical trial is to learn if Autonomic Recalibration works to reduce sympathetic dominance to alleviate dysfunctional myofascial pain. The main questions it aims to answer are:

How is the Autonomic Nervous System (ANS) affected during Autonomic Recalibration Treatment (ART)? How are myofascial tissue properties impacted from ART?

Participants will:

Have 2 treatments of ART on consecutive days. Wear sensors to track HRV (heart rate variability) and GSR to verify autonomic recalibration.

Measure changes in range of motion by wearing a Rokoko motion capture suit. Measure changes in muscle stiffness through shear wave elastography.

DETAILED DESCRIPTION:
Myofascial pain contributes to opioid misuse and opioid use disorder. Alternative non-drug therapies for myofascial pain, such as osteopathic manipulative treatment, are critical areas of research. An unexplored approach in osteopathic manipulative treatment is recruiting the regulatory assistance of the autonomic nervous system (ANS) to alleviate myofascial pain. Autonomic Recalibration Technique (ART) is a manual and behavioral approach that employs osteopathic principles in addressing the neurobiological mechanisms that regulate myofascial pain. Our central hypothesis is that ART utilizes ANS regulation to restore myofascial function and alleviate chronic myofascial pain. The scientific premise of this proposal is the need to document mechanistic evidence that the ANS can be recruited to alleviate and eliminate pain by employing osteopathic principles. While elements of this approach have been employed by various practitioners, including manual and integrative clinicians including osteopaths, the innovation is to combine a manual bottom-up approach to shut down sympathetic tone, and a top-down approach to address trauma-based triggers that propagate pain. If successful, these preclinical data will be used in future grants to propose a clinical trial of ART as an additional technique in osteopathic manipulative treatment to provide an alternative to surgical or drug treatment of chronic myofascial pain.

ELIGIBILITY:
Inclusion Criteria:

* dysfunctional myofascial pain, i.e., ongoing pain not relevant to an acute perturbation (e.g., recent injury) or known underlying condition (e.g., cancer).

Exclusion Criteria:

* known skin allergies to gel as found in common cosmetic or household products
* can't make treatment appointments on two consecutive days
* myofascial pain is deemed functional (normal response to acute injury or ongoing pathology)
* lacking a COVID-19 vaccination and a booster shot.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-04-27 (Actual); Primary Completion 2023-08-24 (Actual); Study Completion 2024-02-27 (Actual)

PRIMARY OUTCOMES:
Pain Intensity (NRS Pain Scale) | Pre/Post for each day of treatment. 2 days total.
  0-10 Pain Rating. 0=no pain to 10=pain as intense as you can imagine
Heart Rate Variability | Pre/Post for each day of treatment. 2 days total.
  Changes in HRV (ms) pre/post and Day 1/Day 2.
Galvanic Skin Response (GSR) | Pre/Post for each day of treatment. 2 days total.
  Comparison of GSR peak counts pre/post and Day 1/Day 2.
Muscle Stiffness using Shear Wave Elastography | Pre/Post for each day of treatment. 2 days total.
  Changes in muscle stiffness (kPa) measured by Ultrasound.
Nociceptive Trigger Points | Pre/Middle/Post for each day of treatment. 2 days total.
  Log of reported trigger points during nociceptive start exam. Taken Pre, Middle, and Post ART on Day 1 and Day 2.
Changes in mobility | Pre/Post for each day of treatment. 2 days total.
  Posture/mobility changes using multivariate morphometric analysis.

CONTACTS AND LOCATIONS:
Overall Officials: William G Pearson, PhD, Principal Investigator — Edward Via College of Osteopathic Medicine, Auburn campus
Locations (1):
- Edward Via College of Osteopathic Medicine, Auburn Campus, Auburn, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Volkow ND, McLellan TA, Cotto JH, Karithanom M, Weiss SR. Characteristics of opioid prescriptions in 2009. JAMA. 2011 Apr 6;305(13):1299-301. doi: 10.1001/jama.2011.401. No abstract available. PMID 21467282
- [Background] Vattigunta S, Weiner S, Nayar SK, Jenkins S, Srikumaran U. Opioid consumption following orthopedic shoulder surgery: a retrospective analysis. J Shoulder Elbow Surg. 2021 Jul;30(7S):S153-S158. doi: 10.1016/j.jse.2021.04.005. Epub 2021 Apr 21. PMID 33892118
- [Background] Turo D, Otto P, Hossain M, Gebreab T, Armstrong K, Rosenberger WF, Shao H, Shah JP, Gerber LH, Sikdar S. Novel Use of Ultrasound Elastography to Quantify Muscle Tissue Changes After Dry Needling of Myofascial Trigger Points in Patients With Chronic Myofascial Pain. J Ultrasound Med. 2015 Dec;34(12):2149-61. doi: 10.7863/ultra.14.08033. Epub 2015 Oct 21. PMID 26491094
- [Background] Reddan MC, Wager TD. Modeling Pain Using fMRI: From Regions to Biomarkers. Neurosci Bull. 2018 Feb;34(1):208-215. doi: 10.1007/s12264-017-0150-1. Epub 2017 Jun 23. PMID 28646349
- [Background] Park G, Kim CW, Park SB, Kim MJ, Jang SH. Reliability and usefulness of the pressure pain threshold measurement in patients with myofascial pain. Ann Rehabil Med. 2011 Jun;35(3):412-7. doi: 10.5535/arm.2011.35.3.412. Epub 2011 Jun 30. PMID 22506152
- [Background] Oliveira-Campelo NM, de Melo CA, Alburquerque-Sendin F, Machado JP. Short- and medium-term effects of manual therapy on cervical active range of motion and pressure pain sensitivity in latent myofascial pain of the upper trapezius muscle: a randomized controlled trial. J Manipulative Physiol Ther. 2013 Jun;36(5):300-9. doi: 10.1016/j.jmpt.2013.04.008. Epub 2013 Jun 12. PMID 23769263
- [Background] Morikawa Y, Takamoto K, Nishimaru H, Taguchi T, Urakawa S, Sakai S, Ono T, Nishijo H. Compression at Myofascial Trigger Point on Chronic Neck Pain Provides Pain Relief through the Prefrontal Cortex and Autonomic Nervous System: A Pilot Study. Front Neurosci. 2017 Apr 11;11:186. doi: 10.3389/fnins.2017.00186. eCollection 2017. PMID 28442987
- [Background] Menendez ME, Ring D, Bateman BT. Preoperative Opioid Misuse is Associated With Increased Morbidity and Mortality After Elective Orthopaedic Surgery. Clin Orthop Relat Res. 2015 Jul;473(7):2402-12. doi: 10.1007/s11999-015-4173-5. Epub 2015 Feb 19. PMID 25694266
- [Background] Mejia-Mejia E, Budidha K, Abay TY, May JM, Kyriacou PA. Heart Rate Variability (HRV) and Pulse Rate Variability (PRV) for the Assessment of Autonomic Responses. Front Physiol. 2020 Jul 23;11:779. doi: 10.3389/fphys.2020.00779. eCollection 2020. PMID 32792970
- [Background] Malliaras P, Rathi S, Burstein F, Watt L, Ridgway J, King C, Warren N. 'Physio's not going to repair a torn tendon': patient decision-making related to surgery for rotator cuff related shoulder pain. Disabil Rehabil. 2022 Jul;44(14):3686-3693. doi: 10.1080/09638288.2021.1879945. Epub 2021 Feb 12. PMID 33577359
- [Background] Maher RM, Hayes DM, Shinohara M. Quantification of dry needling and posture effects on myofascial trigger points using ultrasound shear-wave elastography. Arch Phys Med Rehabil. 2013 Nov;94(11):2146-50. doi: 10.1016/j.apmr.2013.04.021. Epub 2013 May 14. PMID 23684553
- [Background] Lok UW, Huang C, Zhou C, Yang L, Ling W, Tang S, Gong P, Madson TJ, Jensen MA, Gay RE, Chen S. Quantitative Shear Wave Speed Assessment for Muscles With the Diagnosis of Taut Bands and/or Myofascial Trigger Points Using Probe Oscillation Shear Wave Elastography: A Pilot Study. J Ultrasound Med. 2022 Apr;41(4):845-854. doi: 10.1002/jum.15764. Epub 2021 Jun 4. PMID 34085301
- [Background] Lavelle ED, Lavelle W, Smith HS. Myofascial trigger points. Anesthesiol Clin. 2007 Dec;25(4):841-51, vii-iii. doi: 10.1016/j.anclin.2007.07.003. PMID 18054148
- [Background] Lamine H, Bennour S, Laribi M, Romdhane L, Zaghloul S. Evaluation of Calibrated Kinect Gait Kinematics Using a Vicon Motion Capture System. Comput Methods Biomech Biomed Engin. 2017 Oct;20(sup1):111-112. doi: 10.1080/10255842.2017.1382886. No abstract available. PMID 29088586
- [Background] Kunz M, Scharmann S, Hemmeter U, Schepelmann K, Lautenbacher S. The facial expression of pain in patients with dementia. Pain. 2007 Dec 15;133(1-3):221-8. doi: 10.1016/j.pain.2007.09.007. Epub 2007 Oct 18. PMID 17949906
- [Background] Kisilewicz A, Madeleine P, Ignasiak Z, Ciszek B, Kawczynski A, Larsen RG. Eccentric Exercise Reduces Upper Trapezius Muscle Stiffness Assessed by Shear Wave Elastography and Myotonometry. Front Bioeng Biotechnol. 2020 Aug 5;8:928. doi: 10.3389/fbioe.2020.00928. eCollection 2020. PMID 32903634
- [Background] Kim J, Loggia ML, Cahalan CM, Harris RE, Beissner F Dr Phil Nat, Garcia RG, Kim H, Wasan AD, Edwards RR, Napadow V. The somatosensory link in fibromyalgia: functional connectivity of the primary somatosensory cortex is altered by sustained pain and is associated with clinical/autonomic dysfunction. Arthritis Rheumatol. 2015 May;67(5):1395-1405. doi: 10.1002/art.39043. PMID 25622796
- [Background] Hayano J, Yuda E. Pitfalls of assessment of autonomic function by heart rate variability. J Physiol Anthropol. 2019 Mar 13;38(1):3. doi: 10.1186/s40101-019-0193-2. PMID 30867063
- [Background] Hansel A, von Kanel R. The ventro-medial prefrontal cortex: a major link between the autonomic nervous system, regulation of emotion, and stress reactivity? Biopsychosoc Med. 2008 Nov 5;2:21. doi: 10.1186/1751-0759-2-21. PMID 18986513
- [Background] Hansberger BL, Baker RT, May J, Nasypany A. A NOVEL APPROACH TO TREATING PLANTAR FASCIITIS - EFFECTS OF PRIMAL REFLEX RELEASE TECHNIQUE: A CASE SERIES. Int J Sports Phys Ther. 2015 Oct;10(5):690-9. PMID 26491619
- [Background] Han HJ, Labbaf S, Borelli JL, Dutt N, Rahmani AM. Objective stress monitoring based on wearable sensors in everyday settings. J Med Eng Technol. 2020 May;44(4):177-189. doi: 10.1080/03091902.2020.1759707. Epub 2020 Jun 26. PMID 32589065
- [Background] Hallman DM, Ekman AH, Lyskov E. Changes in physical activity and heart rate variability in chronic neck-shoulder pain: monitoring during work and leisure time. Int Arch Occup Environ Health. 2014;87(7):735-44. doi: 10.1007/s00420-013-0917-2. Epub 2013 Oct 26. PMID 24162088
- [Background] Ge HY, Fernandez-de-las-Penas C, Arendt-Nielsen L. Sympathetic facilitation of hyperalgesia evoked from myofascial tender and trigger points in patients with unilateral shoulder pain. Clin Neurophysiol. 2006 Jul;117(7):1545-50. doi: 10.1016/j.clinph.2006.03.026. Epub 2006 Jun 5. PMID 16737848
- [Background] Gandhi RA, Marques JL, Selvarajah D, Emery CJ, Tesfaye S. Painful diabetic neuropathy is associated with greater autonomic dysfunction than painless diabetic neuropathy. Diabetes Care. 2010 Jul;33(7):1585-90. doi: 10.2337/dc09-2314. PMID 20587724
- [Background] Fede C, Petrelli L, Guidolin D, Porzionato A, Pirri C, Fan C, De Caro R, Stecco C. Evidence of a new hidden neural network into deep fasciae. Sci Rep. 2021 Jun 16;11(1):12623. doi: 10.1038/s41598-021-92194-z. PMID 34135423
- [Background] Ertekin E, Kasar ZS, Turkdogan FT. Is early diagnosis of myofascial pain syndrome possible with the detection of latent trigger points by shear wave elastography? Pol J Radiol. 2021 Jul 12;86:e425-e431. doi: 10.5114/pjr.2021.108537. eCollection 2021. PMID 34429789
- [Background] Clar C, Tsertsvadze A, Court R, Hundt GL, Clarke A, Sutcliffe P. Clinical effectiveness of manual therapy for the management of musculoskeletal and non-musculoskeletal conditions: systematic review and update of UK evidence report. Chiropr Man Therap. 2014 Mar 28;22(1):12. doi: 10.1186/2045-709X-22-12. PMID 24679336
- [Background] Charles D, Hudgins T, MacNaughton J, Newman E, Tan J, Wigger M. A systematic review of manual therapy techniques, dry cupping and dry needling in the reduction of myofascial pain and myofascial trigger points. J Bodyw Mov Ther. 2019 Jul;23(3):539-546. doi: 10.1016/j.jbmt.2019.04.001. Epub 2019 Apr 4. PMID 31563367
- [Background] Cederqvist S, Flinkkila T, Sormaala M, Ylinen J, Kautiainen H, Irmola T, Lehtokangas H, Liukkonen J, Pamilo K, Ridanpaa T, Sirnio K, Leppilahti J, Kiviranta I, Paloneva J. Non-surgical and surgical treatments for rotator cuff disease: a pragmatic randomised clinical trial with 2-year follow-up after initial rehabilitation. Ann Rheum Dis. 2021 Jun;80(6):796-802. doi: 10.1136/annrheumdis-2020-219099. Epub 2020 Dec 3. PMID 33272959
- [Background] Cauzzo S, Singh K, Stauder M, Garcia-Gomar MG, Vanello N, Passino C, Staab J, Indovina I, Bianciardi M. Functional connectome of brainstem nuclei involved in autonomic, limbic, pain and sensory processing in living humans from 7 Tesla resting state fMRI. Neuroimage. 2022 Apr 15;250:118925. doi: 10.1016/j.neuroimage.2022.118925. Epub 2022 Jan 21. PMID 35074504
- [Background] Bolanos, L., Vicente, J. M., Vivas, O. A., & Sabater-Navarro, J. M. (2019). Electrodermal activity in relation to diabetes, autonomic neuropathy and aging: a preliminary study. Ingeniería E Investigación, 39(3), 27-33.
- [Background] Babatunde OO, Jordan JL, Van der Windt DA, Hill JC, Foster NE, Protheroe J. Effective treatment options for musculoskeletal pain in primary care: A systematic overview of current evidence. PLoS One. 2017 Jun 22;12(6):e0178621. doi: 10.1371/journal.pone.0178621. eCollection 2017. PMID 28640822
- [Background] Albertin ES, Walters M, May J, Baker RT, Nasypany A, Cheatham S. AN EXPLORATORY CASE SERIES ANALYSIS OF THE USE OF PRIMAL REFLEX RELEASE TECHNIQUE TO IMPROVE SIGNS AND SYMPTOMS OF HAMSTRING STRAIN. Int J Sports Phys Ther. 2020 Apr;15(2):263-273. PMID 32269860